CLINICAL TRIAL: NCT05196269
Title: Comparing Decision on Match of Expectations and Aesthetics Using a Conventional Versus a Cloud-based Healthcare Platform Approach in Breast Cancer Patients Proposed for Locoregional Treatment: A Prospective Randomized Trial
Brief Title: Comparing Decision on Aesthetics After Breast Cancer Locoregional Treatment.
Acronym: CINDERELLA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacao Champalimaud (Other)
Collaborators: European Commission (Other); INESC TEC - Institute for Systems and Computer Engineering, Technology and Science (Porto, Portugal) (Unknown); Cankado GmbH (Industry); FCiências.ID - Associação para a Investigação e Desenvolvimento de Ciências (Lisbon, Portugal) (Unknown); Bocconi University (Other)
Responsible Party: Principal Investigator, Maria-Joao Cardoso, Head Breast Surgeon - MD, PhD, Fundacao Champalimaud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CINDERELLA
Record Dates: First submitted 2021-10-26; First posted 2022-01-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Surgery; Radiation; Artificial Intelligence; Outcomes; Aesthetics; Expectations; Satisfaction; Quality of life; Digital Platform
MeSH Terms: conditions — Breast Neoplasms; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Prospective randomized open trial with parallel groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Artificial Intelligence and Digital Health Arm (Experimental): Using an Artificial Intelligence approach integrated in a cloud-based healthcare platform CANKADO to give the patient complete information about the proposed type of locoregional treatment and access to photographs and data of patients with similar characteristics previously treated with the same technique. All interaction will be through the CANKADO Platform.
  Interventions: Device: Artificial Intelligence and Digital Health Arm
- Control Comparator (Other): The standard approach of proposing patients for locoregional treatment with or without printed or digital materials and hypothetic visualization of results.
  Interventions: Device: Artificial Intelligence and Digital Health Arm

INTERVENTIONS:
Device: Artificial Intelligence and Digital Health Arm — A previous large database repository of images having thousands of pre and postoperative photographs of breast cancer patients proposed for locoregional treatment with clinical and biometric data will be matched using artificial intelligence within the CANKADO platform. Patients proposed for breast cancer locoregional treatment will have access to the software installed, and they will have access to all the information about the type of treatment they will receive. All the questions and questionnaires will be filled out online, and they can visualise the expected outcome from excellent to poor.
  Other Names: Artificial Intelligence and cloud-based digital health platform

SUMMARY:
Breast cancer is the most commonly diagnosed cancer, with an estimated 2.3 million new cases per year globally. Approximately 90% of these patients will undergo breast surgery with/without radiation (locoregional treatment). Different surgical techniques can be offered to the patient, each leading to completely different aesthetic outcomes. Moreover, the aesthetic outcome could be completely different for patients undergoing the same surgery based on individual patient factors (e.g., age, body habitus). In the CINDERELLA trial, the investigators will be using the (Breast Locoregional (BreLO) AI system (an artificial intelligence-based tool for the classification of aesthetic outcomes and matching data and photographs) integrated into CANKADO (a cloud-based healthcare platform) to create an easy-to-use application that can be used on any electronic device, to simulate visually to the patient the aesthetic outcome of a certain surgery or radiation treatment. In the CINDERELLA trial, the investigators plan to compare whether the application helped fulfil the expectations and lead to a better quality of life compared with the classical approach. In the classical approach (control arm), doctors usually propose a locoregional treatment and explain theoretically how the result will be. Nurses help by explaining further details about the surgery and possible outcomes. In most centres, no photographic evaluation is done, and expectations are not measured. The CINDERELLA trial will help overcome miscommunication and potential boundaries in the patient's or physician's understanding of the potential outcomes of locoregional breast cancer treatment.

DETAILED DESCRIPTION:
The CINDERELLA clinical trial will be an open, prospective randomized trial that Champalimaud Foundation will coordinate. Five clinical centres agreed to participate in the trial. The trial will be designed and reported according to the latest SPIRIT-AI and CONSORT-AI guidelines.

The randomization will be made by adopting a dynamical approach following the Minimization Method. Assignment of the recruited patients to the study arms will take into account the stratification of the participants (younger and older than 50 / breast-conserving or mastectomy / mastectomy with or without radiotherapy), aiming to reduce bias and confounding by assuring the balance of the group.

After being proposed to the trial and checked for all the eligibility criteria, patients will be given the complete patient information before signing the informed consent.

For the five centres, a minimum of 515 patients should be enrolled in each arm of the study. After randomization, the patient will either follow:

1. - The intervention arm with the CINDERELLA APProach with the introduction and access to CANKADO with the BreLO AI system. The Expectations Questionnaire, Healthcare Professionals Multidimensional Evaluation Questionnaire and standard patient-reported outcomes measures (PROMs) (EQ-5D-5L and BREAST Q ICHOM) will be filed electronically. Standard photographic capture will be taken at this point. After the photographic capture, the BreLO-AI will match the patient biometrics and images with the more identical case existing in the BreLO repository and already classified by the BCCT.core into excellent, good, fair and poor. The new patient can then visualize the results. In case of doubts, queries will be answered through the app or, if needed, by phone call or booking another appointment. Questionnaires and Photographs will be repeated after wound healing is complete, six months and one year after the end of treatment (surgery or radiotherapy if radiotherapy was done).
2. - The control arm with the Conventional approach with a theoretical explanation by the doctor/nurse of the proposed locoregional treatment and possible outcomes. The Expectations Questionnaire, Healthcare Professionals Multidimensional Evaluation Questionnaire and standard PROMs (EQ-5D-5L and BREAST Q ICHOM) will be filed electronically. Standard photographic capture will be taken at this point. In case of doubts, the patient will book another appointment with the doctor/nurse, as usually done in routine practice. Questionnaires and Photographs will be repeated after healing is complete, six months and one year after the end of treatment (surgery or radiotherapy if radiotherapy was done).

Digital Photography (same protocol for all participating centres) - a similar protocol for image capture will exist for all centres. The standalone photography with an automatic robot will be progressively implemented (www.photorobot.com).

DATA COLLECTION

PATIENT-RELATED FACTORS

* Date of birth, Weight / Height / BMI, Thoracic perimeter, Bra size and cup
* Education degree, Profession, Hobbies
* Marital status, Pregnancies and offspring
* Breast-feeding, Menopausal status
* Smoking
* Connective tissue diseases
* Confirmed Pathogenic Germline Variant

TUMOUR-RELATED FACTORS

* Unilateral (unifocal, multifocal, multicentric) Bilateral
* Histological type according to World Health Organization (WHO) classification (e.g., invasive ductal carcinoma, lobular carcinoma) (size in mm) staging ER, PR, Her2, Ki67, cTNM - pTNM / ypTNM

TREATMENT-RELATED FACTORS

*Type of Surgery/ Type of Reconstruction: (data collection regarding surgery should also include acellular dermal matrice (ADM) if used - type and placement) TYPE OF SURGERY: C1 - Conservative surgery - unilateral or bilateral, C2 - Conservative surgery with bilateral reduction (uni or bilateral), C3 - Conservative surgery with LD or LICAP/TDAP, C4 - Conservative surgery with bilateral breast augmentation, M1 - Mastectomy with unilateral reconstruction with implant, M2 - Mastectomy with unilateral reconstruction with autologous flap, M3 - Mastectomy with bilateral reconstruction with implants, M4 - Mastectomy with bilateral reconstruction with autologous flaps, M5 - Mastectomy with unilateral reconstruction with implant and contralateral symmetrisation with implant (augmentation), M6 - Mastectomy with unilateral reconstruction with implant and contralateral symmetrisation with reduction, M7 - Mastectomy with unilateral reconstruction with autologous flap and contralateral symmetrisation with reduction, M8 - Mastectomy with unilateral reconstruction with autologous flap and contralateral symmetrisation with implant (augmentation).

STATISTICAL ANALYSIS

An extensive descriptive analysis will be performed to characterize the groups in detail and the outcomes of the study at baseline as well as in the following points of data collection. Concerning the primary objectives, models of the class of generalized linear mixed models (in particular, multinomial regression models for ordinal data) will be estimated to evaluate the effect of the training and the women's characteristics on their evaluation of the aesthetic results of the surgery at each time and along time through longitudinal analysis. The Wilcoxon signed rank test for pairs will also be used to evaluate the effect of training on the level of agreement of the expectations and the final result. Weighted Cohen's k will be calculated for both groups (train and control) and compared using a statistical test and/or bootstrap techniques to assess the improvement in the ability to classify the aesthetic result of their surgery provided by training. A measure of similarity between self-evaluation and the BCCT.core will be computed for each participant, and a beta regression model will be estimated to assess the effect of training, controlling variables that can play as confounders, such as women's and disease characteristics at each time point and in a longitudinal perspective. Concerning the secondary objectives, the patient-reported outcome measures administered will be scored according to the official guidelines provided by the developers of the instruments. Besides the descriptive statistics, the outcomes will be compared between groups using adequate statistical tests. Again, models of the class of the general linear mixed models will be used.

ELIGIBILITY:
Inclusion :

* More than 18 years old
* Written informed consent
* Primary breast cancer in situ or invasive without evidence of systemic disease - non Stage IV or locally advanced non-operable breast cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Uni or Bilateral surgery even if prophylactic in one side
* Capacity to use a web-based app autonomously or with home-based support

Exclusion:

* Mastectomy without reconstruction
* Pregnancy or lactation
* Previous radiation to breast/chest (e.g., lymphoma)
* Previous ipsilateral breast surgery due to malignant disease.
* Other neoplasm in the last 5 years (excluding basal cell carcinoma of the skin and adequately treated carcinoma in situ of the cervix)
* Severe skin disease that will contra-indicate the use of radiotherapy
* Prophylactic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The solution we aim to apply in clinical practice is non-sex/gender specific. However, the proposal focuses on breast cancer, where there will be a predominance of female participants.
  The incidence of breast cancer contrasts strikingly according to gender, with approximately 1% of all tumours occurring in males. Although breast conservation can also be offered to men, it is a rare practice, and most men are submitted to mastectomy without breast reconstruction.
  As a consequence, it will be very difficult to recruit male patients to the study and obtain data that will allow any conclusions taking into account that mastectomy without reconstruction is out of our scope, and as such will not be included in our trial.
Enrollment: 1030 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Agreement between patients expectations before and after treatment in both the intervention and the control arm | 12 months after locoregional treatment (surgery or radiotherapy in case adjuvant radiotherapy is done)
  Agreement between patient's expectations about the aesthetic outcome measured before and after treatment, evaluated at 12 months after treatment (Cohen's Kappa and weighted Kappa Statistics) both the intervention and the control arm.
Agreement about the aesthetic outcome between the objective evaluation and self- evaluation measured after treatment in both the intervention and the control arm | 12 months after locoregional treatment (surgery or radiotherapy in case adjuvant radiotherapy is done)
  Agreement about the aesthetic outcome between the AI evaluation tool (BCT.core software) and self- evaluation after treatment (Cohen's Kappa and weighted Kappa Statistics) in both the intervention and the control arm.

SECONDARY OUTCOMES:
Patient's body image satisfaction after surgery measured through the BREAST-Q - International Consortium for Health Outcomes Measurement (ICHOM) questionnaire | 12 months after locoregional treatment (surgery or radiotherapy in case adjuvant radiotherapy is done)
  Body image perception and satisfaction using the BREAST-Q ICHOM questionnaire. The scale scores from 0 lowest to 100 highest (body image satisfaction) in both the intervention and the control arm.
Resource consumption a) time spent in hospital b) number of appointments c) duration until treatment d) out of pocket expenditure, additional care sought by patients | 12 months after locoregional treatment (surgery or radiotherapy in case adjuvant radiotherapy is done
  Resource consumption (cost per patient evaluated by the amount of appointments between the surgical proposal by the surgeon and the end of the trial) in both the intervention and control arm.
Patient's general health-related quality of life evaluated in both the intervention and control arm with the EQ-5D-5L questionnaire | 12 months after locoregional treatment (surgery or radiotherapy in case adjuvant radiotherapy is done)
  How results impact in patients general quality of life evaluated in both the intervention and control arm with the EQ-5D-5L questionnaire. The scale scores from 0 lowest to 100 highest. A high scale score represents a high/healthy level of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Joao Cardoso, MD, PhD, Principal Investigator — Champalimaud Foundation
Locations (6):
- Universitätsklinikum Heidelberg, Heidelberg, Germany
- Sheba Medical Center, Ramat Gan, Israel
- IRCCS Ospedale San Raffaele, Milan, Italy
- Poland (2):
  - Copernicus Mamma Centrum, Wojewodzkie Centrum Onkologii, Copernicus Podmiot Leczniczy, Gdansk, Pomeranian
  - Gdański Uniwersytet Medyczny, Gdansk, Pomeranian
- Champalimaud Research and Clinical Centre, Champalimaud Foundation, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pilleron S, Soto-Perez-de-Celis E, Vignat J, Ferlay J, Soerjomataram I, Bray F, Sarfati D. Estimated global cancer incidence in the oldest adults in 2018 and projections to 2050. Int J Cancer. 2021 Feb 1;148(3):601-608. doi: 10.1002/ijc.33232. Epub 2020 Aug 17. PMID 32706917
- [Background] Kim MK, Kim T, Moon HG, Jin US, Kim K, Kim J, Lee JW, Kim J, Lee E, Yoo TK, Noh DY, Minn KW, Han W. Effect of cosmetic outcome on quality of life after breast cancer surgery. Eur J Surg Oncol. 2015 Mar;41(3):426-32. doi: 10.1016/j.ejso.2014.12.002. Epub 2014 Dec 19. PMID 25578249
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Background] Zehra S, Doyle F, Barry M, Walsh S, Kell MR. Health-related quality of life following breast reconstruction compared to total mastectomy and breast-conserving surgery among breast cancer survivors: a systematic review and meta-analysis. Breast Cancer. 2020 Jul;27(4):534-566. doi: 10.1007/s12282-020-01076-1. Epub 2020 Mar 12. PMID 32162181
- [Background] Harris JR, Levene MB, Svensson G, Hellman S. Analysis of cosmetic results following primary radiation therapy for stages I and II carcinoma of the breast. Int J Radiat Oncol Biol Phys. 1979 Feb;5(2):257-61. doi: 10.1016/0360-3016(79)90729-6. No abstract available. PMID 110740
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Ong WL, Schouwenburg MG, van Bommel ACM, Stowell C, Allison KH, Benn KE, Browne JP, Cooter RD, Delaney GP, Duhoux FP, Ganz PA, Hancock P, Jagsi R, Knaul FM, Knip AM, Koppert LB, Kuerer HM, McLaughin S, Mureau MAM, Partridge AH, Reid DP, Sheeran L, Smith TJ, Stoutjesdijk MJ, Vrancken Peeters MJTFD, Wengstrom Y, Yip CH, Saunders C. A Standard Set of Value-Based Patient-Centered Outcomes for Breast Cancer: The International Consortium for Health Outcomes Measurement (ICHOM) Initiative. JAMA Oncol. 2017 May 1;3(5):677-685. doi: 10.1001/jamaoncol.2016.4851. PMID 28033439
- [Background] Ciani O, Federici CB. Value Lies in the Eye of the Patients: The Why, What, and How of Patient-reported Outcomes Measures. Clin Ther. 2020 Jan;42(1):25-33. doi: 10.1016/j.clinthera.2019.11.016. Epub 2020 Jan 10. PMID 31932079
- [Background] Fitzal F, Krois W, Trischler H, Wutzel L, Riedl O, Kuhbelbock U, Wintersteiner B, Cardoso MJ, Dubsky P, Gnant M, Jakesz R, Wild T. The use of a breast symmetry index for objective evaluation of breast cosmesis. Breast. 2007 Aug;16(4):429-35. doi: 10.1016/j.breast.2007.01.013. Epub 2007 Mar 26. PMID 17382546
- [Background] Cardoso MJ, Cardoso J, Amaral N, Azevedo I, Barreau L, Bernardo M, Christie D, Costa S, Fitzal F, Fougo JL, Johansen J, Macmillan D, Mano MP, Regolo L, Rosa J, Teixeira L, Vrieling C. Turning subjective into objective: the BCCT.core software for evaluation of cosmetic results in breast cancer conservative treatment. Breast. 2007 Oct;16(5):456-61. doi: 10.1016/j.breast.2007.05.002. Epub 2007 Jul 2. PMID 17606373
- [Background] Cardoso JS, Cardoso MJ. Towards an intelligent medical system for the aesthetic evaluation of breast cancer conservative treatment. Artif Intell Med. 2007 Jun;40(2):115-26. doi: 10.1016/j.artmed.2007.02.007. Epub 2007 Apr 8. PMID 17420117
- [Background] Heil J, Dahlkamp J, Golatta M, Rom J, Domschke C, Rauch G, Cardoso MJ, Sohn C. Aesthetics in breast conserving therapy: do objectively measured results match patients' evaluations? Ann Surg Oncol. 2011 Jan;18(1):134-8. doi: 10.1245/s10434-010-1252-4. Epub 2010 Aug 10. PMID 20697820
- [Background] Cardoso MJ, Cardoso JS, Oliveira HP, Gouveia P. The breast cancer conservative treatment. Cosmetic results - BCCT.core - Software for objective assessment of esthetic outcome in breast cancer conservative treatment: A narrative review. Comput Methods Programs Biomed. 2016 Apr;126:154-9. doi: 10.1016/j.cmpb.2015.11.010. Epub 2015 Dec 9. PMID 26707372
- [Background] Cardoso JS, Silva W, Cardoso MJ. Evolution, current challenges, and future possibilities in the objective assessment of aesthetic outcome of breast cancer locoregional treatment. Breast. 2020 Feb;49:123-130. doi: 10.1016/j.breast.2019.11.006. Epub 2019 Nov 21. PMID 31790958
- [Background] Ciani O, Salcher-Konrad M, Meregaglia M, Smith K, Gorst SL, Dodd S, Williamson PR, Fattore G. Patient-reported outcome measures in core outcome sets targeted overlapping domains but through different instruments. J Clin Epidemiol. 2021 Aug;136:26-36. doi: 10.1016/j.jclinepi.2021.03.003. Epub 2021 Mar 6. PMID 33689837
- [Background] van Egdom LSE, Pusic A, Verhoef C, Hazelzet JA, Koppert LB. Machine learning with PROs in breast cancer surgery; caution: Collecting PROs at baseline is crucial. Breast J. 2020 Jun;26(6):1213-1215. doi: 10.1111/tbj.13804. Epub 2020 Mar 11. PMID 32160651
- [Background] Pfob A, Sidey-Gibbons C, Schuessler M, Lu SC, Xu C, Dubsky P, Golatta M, Heil J. Contrast of Digital and Health Literacy Between IT and Health Care Specialists Highlights the Importance of Multidisciplinary Teams for Digital Health-A Pilot Study. JCO Clin Cancer Inform. 2021 Jun;5:734-745. doi: 10.1200/CCI.21.00032. PMID 34236897
- [Background] Brunet J, Price J. A scoping review of measures used to assess body image in women with breast cancer. Psychooncology. 2021 May;30(5):669-680. doi: 10.1002/pon.5619. Epub 2021 Jan 21. PMID 33480160
- [Background] Flitcroft K, Brennan M, Spillane A. Women's expectations of breast reconstruction following mastectomy for breast cancer: a systematic review. Support Care Cancer. 2017 Aug;25(8):2631-2661. doi: 10.1007/s00520-017-3712-x. Epub 2017 May 4. PMID 28474240
- [Background] Fuzesi S, Becetti K, Klassen AF, Gemignani ML, Pusic AL. Expectations of breast-conserving therapy: a qualitative study. J Patient Rep Outcomes. 2019 Dec 27;3(1):73. doi: 10.1186/s41687-019-0167-5. PMID 31883052
- [Background] Biganzoli L, Marotti L, Hart CD, Cataliotti L, Cutuli B, Kuhn T, Mansel RE, Ponti A, Poortmans P, Regitnig P, van der Hage JA, Wengstrom Y, Rosselli Del Turco M. Quality indicators in breast cancer care: An update from the EUSOMA working group. Eur J Cancer. 2017 Nov;86:59-81. doi: 10.1016/j.ejca.2017.08.017. Epub 2017 Sep 28. PMID 28963914
- [Background] Cano SJ, Klassen AF, Scott AM, Pusic AL. A closer look at the BREAST-Q((c)). Clin Plast Surg. 2013 Apr;40(2):287-96. doi: 10.1016/j.cps.2012.12.002. PMID 23506769
- [Background] Preuss J, Lester L, Saunders C. BCCT.core - can a computer program be used for the assessment of aesthetic outcome after breast reconstructive surgery? Breast. 2012 Aug;21(4):597-600. doi: 10.1016/j.breast.2012.05.012. Epub 2012 Jun 17. PMID 22709973
- [Background] Berger VW, Bour LJ, Carter K, Chipman JJ, Everett CC, Heussen N, Hewitt C, Hilgers RD, Luo YA, Renteria J, Ryeznik Y, Sverdlov O, Uschner D; Randomization Innovative Design Scientific Working Group. A roadmap to using randomization in clinical trials. BMC Med Res Methodol. 2021 Aug 16;21(1):168. doi: 10.1186/s12874-021-01303-z. PMID 34399696
- [Derived] Borsoi L, Listorti E, Ciani O; CINDERELLA Consortium. Artificial-Intelligence Cloud-Based Platform to Support Shared Decision-Making in the Locoregional Treatment of Breast Cancer: Protocol for a Multidimensional Evaluation Embedded in the CINDERELLA Clinical Trial. Pharmacoecon Open. 2024 Nov;8(6):945-959. doi: 10.1007/s41669-024-00519-1. Epub 2024 Sep 12. PMID 39264499